CLINICAL TRIAL: NCT04772495
Title: The Potential Candidate miRNA Biomarkers in Multiple Sclerosis
Brief Title: miRNA Biomarkers in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Şenay Görücü Yılmaz, Assoc. Prof., University of Gaziantep
Other Study IDs: 2015/7
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis; miRNA; Epigenetic; Biomarker
Keywords: Multiple sclerosis; miRNA biomarkers; peripheral blood molecular diagnostics
MeSH Terms: conditions — Multiple Sclerosis | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: with Multiple sclerosis
  Interventions: Genetic: miRNA
- Control group: not Multiple sclerosis
  Interventions: Genetic: miRNA

INTERVENTIONS:
Genetic: miRNA — miRNA effect on Multiple sclerosis pathology

SUMMARY:
Multiple Sclerosis (MS) characterized by demyelination and axonal degeneration is a chronic inflammatory disease of the central nervous system (CNS). Recent studies have shown that dysregulated miRNAs alter immune responses, so they may have roles basis on various genetic diseases such as MS and may be potential targets for biomarkers and new therapeutic approaches. In this study, we evaluated the dysregulation of miRNA expression levels at MS and MS stages. We also discussed the potential of these miRNAs to be biomarkers and/or therapeutic targets in MS.

ELIGIBILITY:
Inclusion Criteria:

* The age of 25 years and above
* at least one Central Nervous System (CNS) demyelination event

Exclusion Criteria:

* with genetic diseases, hypertension, head trauma, neuropsychiatric disease, diabetes mellitus, hypertension, cardiac failure, hepatic failure, renal failure, Thalassemia, Sickle cell disease, iron deficiency, and B12 deficiency

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who had been diagnosed with Multiple sclerosis and healthy male and female
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
miRNA expression | intraoperative
  peripheral blood miRNA expressions

IPD SHARING:
Plan to Share IPD: Undecided